CLINICAL TRIAL: NCT01078883
Title: Association Between Respiratory Muscle Performance and Functional Capacity in Patients With Primary Stage IIIb & IV Lung Cancer
Brief Title: Respiratory Muscle Performance and Functional Capacity in Primary Stage IIIb and IV Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chung-Chun Lai, Physical Therapy Center, National Taiwan University Hospital
Other Study IDs: 20090805R
Record Dates: First submitted 2010-02-28; First posted 2010-03-02 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-12

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Respiratory muscle strength; Dyspnea; Functional capacity
MeSH Terms: conditions — Lung Neoplasms; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung cancer: Patients with primary stage IIIb and IV lung cancer

SUMMARY:
The purpose of our study is to investigate the association between respiratory muscle performance, functional capacity, dyspnea, anxiety/depression symptom, 1-year respiratory morbidity rate, and 1-year mortality in patients with primary stage IIIb and IV lung cancer.

DETAILED DESCRIPTION:
Background and Purpose: Respiratory muscle function is important in sustaining the levels of physical activity required for daily life. The purpose of our study is to investigate the association between respiratory muscle performance, functional capacity, dyspnea, anxiety/depression symptom, 1-year respiratory morbidity rate, and 1-year mortality in patients with primary stage IIIb and IV lung cancer.

Methods: A total of 120 patients with newly diagnosed primary stage IIIb and IV lung cancer will be recruited from the National Taiwan University Hospital. Demographic and clinical signs/syndromes will be obtained from the chart. Pain and dyspnea will be measured using visual analog scale. Respiratory muscle strength will be tested by measuring maximal inspiratory and expiratory pressure (PImax and PEmax, respectively). Spirometric variables, forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) will be measured. Functional capacity will be measured using Karnofsky performance status and Simmonds functional assessment. Anxiety/depression symptom will be measured using Hospital Anxiety and Depression Scale. One year respiratory complication morbidity and 1-year mortality will be recorded in prospective nature. Spearman's and Pearson correlation coefficient will be used to test the relationship between respiratory muscle performance and multiple variables. Univariate and stepwise multiple regression analyses will be used to identify factors associated with respiratory muscle performance, functional capacity, one-year respiratory morbidity and one-year mortality rate in patients with primary stage IIIb and IV lung cancer.

Clinical relevance: The prevalence of lung cancer is increasing in the recent years. The attempt to understand the relations between respiratory muscle performance, functional capacity and associated clinical courses will shed light on whether chest physical therapy intervention will be beneficial for patients with primary IIIb and IV lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stage IIIb/V lung cancer
* Normal cognition (a Mini Mental State Examination score of more than/equal to 24 points)
* Able to finish all tests

Exclusion Criteria:

* A clinical diagnosis affecting respiratory muscle function and functional activity performance (e.g. acute pneumonia)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary stage IIIb and IV lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
1-year respiratory morbidity rate and 1-year mortality rate | 1 year

SECONDARY OUTCOMES:
respiratory muscle performance, functional capacity, dyspnea, anxiety/depression symptom | 1-2 days

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Chun Lai, MS., Principal Investigator — Physical Thaerapy Center, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan